## **Chronic Liver Disease in Urea Cycle Disorders**

ClinicalTrials.gov Identifier: NCT03721367

5-11-2022

Demographic characteristics, medical history, and liver biomarkers were summarized usingmeans and standard deviations for continuous outcomes and counts and frequencies for categorical outcomes. For each outcome, we stratified subject characteristics summaries by normal or abnormal readings. For the strength of association between outcome measures and subject characteristics, univariate analyses were used (independent t-test for comparison of means and chi-square test for comparison of proportions). P < 0.05 (nominal) was considered as statistically significant. All statistical analyses were conducted using R or Graphpad Prism v.8.4.2 software (San Diego, CA).